CLINICAL TRIAL: NCT01256086
Title: Relative Potency of Formoterol Novolizer® 12 µg Compared to Formoterol Aerolizer® 12 µg in Patients With Stable Asthma Using Bronchoprovocation With Methacholine as a Bioassay Randomized, Double-blind, Four-period, Four-sequence Cross-over Trial
Brief Title: Relative Potency of Formoterol Novolizer® 12 µg Compared to Formoterol Aerolizer® 12 µg
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MEDA Pharma GmbH & Co. KG (Industry)
Collaborators: ClinResearch, GmbH (Other); Trio Clinical Research, LLC, Raleigh, USA (Unknown); NuCara Pharmacy, Waterloo, USA (Unknown); Prof. Hochhaus, Gainesville, USA (Unknown)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D-64428-3278; IND #101,246 (Registry Identifier: IND #101,246)
Record Dates: First submitted 2010-12-07; First posted 2010-12-08 (Estimated); Results first posted 2012-09-12 (Estimated); Last update posted 2022-02-11 (Actual); Status verified 2012-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 24 µg Formoterol Novolizer (Experimental): 12µg Formoterol Novolizer#1 + 12µg Formoterol Novolizer#2 + Placebo Aerolizer#1 + Placebo Aerolizer #2
  Interventions: Drug: Formatris 24µg
- 12µg Formoterol Novolizer (Experimental): 12µg Formoterol Novolizer#1 + Placebo Novolizer#2 + Placebo Aerolizer#1 + Placebo Aerolizer #2
  Interventions: Drug: Formatris 12µg
- 24 µg Formoterol Aerolizer (Active Comparator): Placebo Novolizer#1 + Placebo Novolizer#2 + 12µg Formoterol Aerolizer#1 + 12µg Formoterol Aerolizer #2
  Interventions: Drug: Foradil P 24µg
- 12µg Formoterol Aerolizer (Active Comparator): Placebo Novolizer#1 + Placebo Novolizer#2 + 12µg Formoterol Aerolizer#1 + Placebo Aerolizer #2
  Interventions: Drug: Foradil P 12µg

INTERVENTIONS:
Drug: Formatris 24µg — 12µg Formoterol Novolizer#1 + 12µg Formoterol Novolizer#2 + Placebo Aerolizer#1 + Placebo Aerolizer #2
  Arms: 24 µg Formoterol Novolizer
Drug: Formatris 12µg — 12µg Formoterol Novolizer#1 + Placebo Novolizer#2 + Placebo Aerolizer#1 + Placebo Aerolizer #2
  Arms: 12µg Formoterol Novolizer
Drug: Foradil P 24µg — Placebo Novolizer#1 + Placebo Novolizer#2 + 12µg Formoterol Aerolizer#1 + 12µg Formoterol Aerolizer #2
  Arms: 24 µg Formoterol Aerolizer
Drug: Foradil P 12µg — Placebo Novolizer#1 + Placebo Novolizer#2 + 12µg Formoterol Aerolizer#1 + Placebo Aerolizer #2
  Arms: 12µg Formoterol Aerolizer

SUMMARY:
The purpose of this study is to estimate the relative potency for bronchoprotective effect of formoterol Novolizer 12 µg (test) compared to formoterol Aerolizer 12 µg (reference).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged from 18 to 60 years (inclusive).
2. Patients with asthma indicated by

   * history of asthma symptoms and
   * airway hyperresponsiveness to methacholine with a provocation concentration of methacholine that cause a 20% decrease in FEV1 (PC20) ≤8 mg/ml at Visit 1.
3. Patients with stable asthma condition with baseline forced expiratory volume in the first second (FEV1) ≥70% predicted at first visit.
4. The PC20 methacholine should increase at least 4-fold after inhaling 24 μg of formoterol Aerolizer (2 applications of 12 μg) at Visit 2.
5. Able to be taught correct inhalation technique for both devices at screening.

Exclusion Criteria:

1. Known hypersensitivity to formoterol, lactose, or methacholine.
2. History of life-threatening asthma in the last three years.
3. Major malignancies including pheochromocytoma within the last 5 years. Exception will be considered where malignancies have been resolved as judged by investigator.
4. Pregnancy, breast-feeding, planned pregnancy during the study, or women of child-bearing potential not using adequate contraception. These methods include total abstinence (no sexual intercourse), oral contraceptives, an intrauterine device (IUD), an etonogestrel implant (Implanon), or medroxyprogesterone acetate injections (Depo-Provera shots). If one of these cannot be used, using contraceptive foam and a condom are recommended.

   Lack of suitability for the study:
5. Screening visit 2 has to be postponed repeatedly.
6. Evidence of respiratory tract infection within 4 weeks before the study (screening visit 1).
7. Seasonal or episodic exposure to an allergen or occupational chemical sensitizer which are likely to vary in symptom presentation and severity during the course of the study (e.g. ragweed sensitive patients in Iowa during Aug-Oct). This does not apply to patients who can be well controlled on therapy.
8. History of non-reversible pulmonary disease; chronic obstructive pulmonary disease (COPD), cystic fibrosis, bronchiectasis, or pulmonary fibrosis.
9. History of severe cardiovascular, renal, neurologic, liver or endocrine dysfunction (patients with well-controlled hypertension, hypercholesterolemia, thyroid disease or diabetes may be included if medication for these diseases does not affect methacholine challenge or formoterol metabolism).
10. History of hemophilia or coagulation disease.
11. Electrocardiogram (ECG) abnormalities of clinical relevance, in particular abnormal prolongation of QT-interval (QTc according to Bazett in women ≥450 msec, in men ≥430 msec).
12. Potassium level below lower limit of laboratory normal range plus 0.3 mmol/l as safety margin.
13. Exacerbation of bronchial asthma requiring emergency department visit or hospitalization during the last 3 months prior to this study.
14. Prior or concomitant treatment with systemic glucocorticosteroids during the last 3 months (a short course of oral corticosteroids for asthma is permissible if for <10 days and at least 30 days have passed).
15. Use of long-acting ß2-agonists in last 3 weeks before the first methacholine challenge or during the study
16. Change in dosage of other controller therapy (inhaled glucocorticosteroids, leukotriene modifier, slow-release theophylline) during the last 3 weeks before the first methacholine challenge or during the study.
17. Use of short-acting ß2-agonists more than thrice a week in the previous month.
18. Inability to temporary withhold the following medications/substances before lung function test:

    * short-acting ß2-agonists and short-acting anticholinergics at least 6 hours,
    * regular long-acting ß2-agonists at least 3 weeks,
    * long-acting anticholinergics at least 36 hours,
    * inhaled glucocorticosteroids at least 2 hours
    * Disodium cromoglycate (DSCG) at least 24 hours,
    * slow release theophylline at least 48 hours,
    * rapid release theophylline at least 24 hours,
    * caffeine at least 4 hours
19. Patients with aspirin induced bronchospasm.
20. Any treatment with ß2-antagonists (including eye drops).
21. Non-cooperative patients, inability to perform outcome measurement correctly.
22. Inability to measure PC20 methacholine after 24 μg of formoterol Aerolizer (PC20 >128 mg/ml).
23. Current smokers or regular smokers during last 12 months or more than 10 pack-year history.
24. Drug or alcohol abuse which would interfere with the patient's proper completion of the protocol assignment.

    Administrative reasons:
25. Participation in another clinical study within 1 month prior to or during this study
26. Lack of ability or willingness to give informed consent.
27. Lack of willingness to have personal study related data collected, archived or transmitted according to protocol.
28. Personnel involved in the planning or conduct of the study.
29. Anticipated non-availability for study visits/procedures.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2010-12; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Hendeles, Professor, Principal Investigator — University of Florida, Gainesville, USA
Locations (3):
- United States (3):
  - University of Florida, Gainesville, Florida
  - University of Iowa, Iowa City, Iowa
  - University of Wisconsin, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient was enrolled in December 2010, last patient completed in July 2011
Pre-assignment Details: During screening phase (within 14 days before but at latest 2 days before randomisation), 2 methacholine tests on separate days (with and without pre-medication) were performed to check the suitability of the patients.
Groups:
- N1A2A1N2: Treatment sequence 12 µg Novolizer - 24 µg Aerolizer - 12 µg Aerolizer - 24 µg Novolizer
- A1N1N2A2: Treatment sequence 12 µg Aerolizer - 12 µg Novolizer - 24 µg Novolizer - 24 µg Aerolizer
- N2A1A2N1: Treatment sequence 24 µg Novolizer - 12 µg Aerolizer - 24 µg Aerolizer - 12 µg Novolizer
- A2N2N1A1: Treatment sequence 24 µg Aerolizer - 24 µg Novolizer - 12 µg Novolizer - 12 µg Aerolizer
Period: Treatment Day 1
Arm/Group | N1A2A1N2 | A1N1N2A2 | N2A1A2N1 | A2N2N1A1
Started | 11 | 11 | 11 | 11
Completed | 11 | 11 | 11 | 11
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Day 2
Arm/Group | N1A2A1N2 | A1N1N2A2 | N2A1A2N1 | A2N2N1A1
Started | 11 | 10 | 9 | 11
Completed | 11 | 10 | 9 | 11
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Day 3
Arm/Group | N1A2A1N2 | A1N1N2A2 | N2A1A2N1 | A2N2N1A1
Started | 11 | 10 | 9 | 11
Completed | 11 | 10 | 9 | 11
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Day 4
Arm/Group | N1A2A1N2 | A1N1N2A2 | N2A1A2N1 | A2N2N1A1
Started | 11 | 10 | 9 | 11
Completed | 11 | 10 | 9 | 11
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- N1A2A1N2: Sequence 1: N1A2A1N2 (Treatment day 1 to treatment day 4) N1 = 12µg Novolizer N2 = 24µg Novolizer A1 = 12µg Aerolizer A2 = 24µg Aerolizer
- A1N1N2A2: Sequence 2: A1N1N2A2 (Treatment day 1 to treatment day 4) N1 = 12µg Novolizer N2 = 24µg Novolizer A1 = 12µg Aerolizer A2 = 24µg Aerolizer
- N2A1A2N1: Sequence 3: N2A1A2N1 (Treatment day 1 to treatment day 4) N1 = 12µg Novolizer N2 = 24µg Novolizer A1 = 12µg Aerolizer A2 = 24µg Aerolizer
- A2N2N1A1: Sequence 4: A2N2N1A1 (Treatment day 1 to treatment day 4) N1 = 12µg Novolizer N2 = 24µg Novolizer A1 = 12µg Aerolizer A2 = 24µg Aerolizer
- Total: Total of all reporting groups
Arm/Group | N1A2A1N2 | A1N1N2A2 | N2A1A2N1 | A2N2N1A1 | Total
Number analyzed (Participants) | 11 | 11 | 11 | 11 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 11 | 11 | 44
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (12) | 35 (13) | 26 (10) | 28 (11) | 30 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 9 | 7 | 31
  Male | 4 | 3 | 2 | 4 | 13
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 11 | 11 | 44

OUTCOME MEASURES:

1. Primary Outcome: PC20 = Provocation Concentration of Methacholine That Cause a 20% Decrease in Forced Expiratory Volume in the First Second (FEV1)
Description: The primary variable is the methacholine PC20 after inhalation of study medication; the PC20 is the concentration of methacholine that - despite protection by study medication - causes a 20% fall in FEV1 compared to the pre-methacholine (post-saline) level of the given study day.
Time Frame: 60 min after application of study medication
Population: Per Protocol Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/ml
Arm/Group | 24 µg Formoterol Novolizer | 12µg Formoterol Novolizer | 24 µg Formoterol Aerolizer | 12µg Formoterol Aerolizer
Number analyzed (Participants) | 38 | 38 | 38 | 38
mg/ml | 35.0 (138.8) | 20.9 (130.1) | 33.2 (96.4) | 17.8 (172.2)
Statistical Analysis 1: Comparison: 24 µg Formoterol Novolizer vs 12µg Formoterol Novolizer vs 24 µg Formoterol Aerolizer vs 12µg Formoterol Aerolizer; Test type: Non-Inferiority or Equivalence — Relative potency of Novolizer compared to Aerolizer. Equivalence was to be concluded if the CI for the relative potency was completely covered by the interval (0.67, 1.50) according to OIP Guideline; Relative potency = 1.13, 90% CI 2-sided [0.94 to 1.38] — Fieller confidence interval for logarithm of relative potency

ADVERSE EVENTS:
Arm/Group | 24 µg Formoterol Novolizer | 12µg Formoterol Novolizer | 24 µg Formoterol Aerolizer | 12µg Formoterol Aerolizer
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/41 | 0/41 | 1/42
Other Adverse Events (participants affected / at risk) | 0/43 | 0/41 | 0/41 | 2/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 24 µg Formoterol Novolizer (N=43) | 12µg Formoterol Novolizer (N=41) | 24 µg Formoterol Aerolizer (N=41) | 12µg Formoterol Aerolizer (N=42)
laryngeal cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Squamous cell carcinoma in situ of the left vocal cord was reported in a female patient with an ongoing history of worsening of vocal hoarseness since 2008. This event was assessed as unlikely related to the use of study drug (Aerolizer 12 µg)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 24 µg Formoterol Novolizer (N=43) | 12µg Formoterol Novolizer (N=41) | 24 µg Formoterol Aerolizer (N=41) | 12µg Formoterol Aerolizer (N=42)
upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — allergic reaction to a cat

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
INSTITUTION shall have the right to publish the results of its part of the study either independently or in collaboration with SPONSOR.In either case, INSTITUTION agrees to submit a copy of any manuscript and/or abstract to SPONSOR for review and comment sixty (60) days prior to its submission for publication. SPONSOR shall have said sixty (60) day period to respond to INSTITUTION with any requested revisions. INSTITUTION agrees to delete information identified by SPONSOR as confidential.